CLINICAL TRIAL: NCT05377359
Title: Lab Evaluation of Novel Hearing Aid Coupling Method
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Collaborators: Sonova Canada Inc. (Industry); Western University, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRF-1082
Record Dates: First submitted 2022-05-11; First posted 2022-05-17 (Actual); Results first posted 2025-03-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-02

CONDITIONS: Hearing Loss
Keywords: Hearing Loss; Hearing Aids; Hearing Aid Receivers
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Intervention Model Description: A single cohort of participants will receive and be assessed in all treatment/intervention conditions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants with Hearing Loss (Experimental): Individuals with hearing loss that meet the candidacy to wear hearing aids with various coupling methods. All interventions are associated with the fitting of binaural hearing aids with various coupling methods. All participants will be assessed under all interventions.
  Interventions: Device: Recordings of Hearing Aids with Open Domes; Device: Recordings of Hearing Aids with Closed Domes; Device: Recordings of Hearing Aids with Novel State 1; Device: Recordings of Hearing Aids with Novel State 2

INTERVENTIONS:
Device: Recordings of Hearing Aids with Open Domes — Receiver-in-the-Canal hearing aids will be used which are programmed to the participant's hearing loss and will be coupled to open domes. Recordings will be made of hearing aid output on a head and torso simulator and played back to participants over headphones.
Device: Recordings of Hearing Aids with Closed Domes — Receiver-in-the-Canal hearing aids will be used which are programmed to the participant's hearing loss and will be coupled with closed domes. Recordings will be made of hearing aid output on a head and torso simulator and played back to participants over headphones.
Device: Recordings of Hearing Aids with Novel State 1 — Receiver-in-the-Canal hearing aids will be used which are programmed to the participant's hearing loss and will be coupled with the new coupling method in its first state. Recordings will be made of hearing aid output on a head and torso simulator and played back to participants over headphones.
Device: Recordings of Hearing Aids with Novel State 2 — Receiver-in-the-Canal hearing aids will be used which are programmed to the participant's hearing loss and will be coupled with the new coupling method in its second state. Recordings will be made of hearing aid output on a head and torso simulator and played back to participants over headphones.

SUMMARY:
Evaluation of different hearing aid coupling methods including two states of a novel coupling method and two traditional coupling methods.

DETAILED DESCRIPTION:
An important decision in the fitting of hearing aids is the selection of the coupling method. Examples of coupling options include universal rubber domes and custom earmolds. When selecting a coupling method, the degree of venting must be considered.

Venting refers to an opening in the coupling method to allow for the sound transmission from the tympanic membrane to the external environment. The degree of venting has a significant impact on the hearing aid user's experience. More closed (or more occluded) coupling means the vent is smaller or non-existent. Occluded fittings allow for more low-frequency amplification, which improves hearing aid performance like directionality, noise reduction and streaming sound quality. However, occluded fittings lead to complaints of the occlusion effect, in which users complain of their own voice as sounding "boomy" and can also lead to a build-up of pressure in the ear canal which users may find uncomfortable. To relieve the occlusion effect and pressure build-ups, more vented (sometimes called open) couplings can be used by allowing low-frequency sounds to leave the ear. Despite a degradation in hearing aid outcomes like directionality, noise reduction and streaming sound quality, open fits are typically preferred for speech quality and own-voice perception - at least for hearing aid users with milder losses and near-normal thresholds at low frequencies.

The fact that two coupling options are associated with two different outcomes means that hearing aid practitioners need to make an important trade-off. Either their patient will enjoy the full breadth of the hearing aid's signal processing potential (via a more occluded fit) or their patient will enjoy better own-voice perception and relief of air pressure in the ear canal(via a more open fit). A coupling method that allows for the best of both options is left to be desired.

A recent development in coupling methods has allowed us to take advantage of both open and closed fittings in a single solution. More occluded coupling allows for more low-frequency amplification which improves hearing aid performance in areas such as directionality, noise reduction, and streaming sound quality. Whereas, open coupling options reduces complaints of the occlusion effect and is preferred for speech quality and own-voice perception by hearing aid users with milder losses. This novel coupling method will function as both an open and closed fitting depending on the environment the listener is in. State 1 is dedicated to loud environments where the listener can take advantage of noise management solutions and for streaming so they can enjoy better sound quality. State 2 is dedicated to quieter environments where the listener can enjoy better physical comfort and own-voice naturality.

This novel coupling method should theoretically exploit the benefits of both open and closed coupling methods. This study is designed to see how this novel coupling method compares to traditional domes and how this coupling method performs in various listening situations.

ELIGIBILITY:
Inclusion Criteria:

* Hearing aid candidate
* Meets the fitting requirements for novel and traditional coupling options
* Healthy outer ear - no visible congenital or traumatic deformity
* Symmetrical hearing loss
* No air-bone gap greater than 10 dB at 500, 1000, 2000, and 4000 Hz
* Ability to answer questions and repeat sentences
* No history of problematic tinnitus or pain/discomfort from loud sounds
* No history of active drainage from the ears in the past 90 days
* Informed consent as documented by signature.

Exclusion Criteria:

* Limited mobility (not able to attend scheduled visits)
* Inability to produce reliable hearing test results
* History of active drainage from the ear in the previous 90 days
* Abnormal appearance of the eardrum and ear canal
* Known psychological problems.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-02-07 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jinyu Qian, PhD, Principal Investigator — Sonova AG
Locations (1):
- Western University - National Centre for Audiology, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Voss SC, Pichora-Fuller MK, Ishida I, Pereira A, Seiter J, El Guindi N, Kuehnel V, Qian J. Evaluating the benefit of hearing aids with motion-based beamformer adaptation in a real-world setup. Int J Audiol. 2022 Aug;61(8):642-654. doi: 10.1080/14992027.2021.1948120. Epub 2021 Aug 7. PMID 34369262
- [Background] Kuk F, Keenan D, Lau CC. Vent configurations on subjective and objective occlusion effect. J Am Acad Audiol. 2005 Oct;16(9):747-62. doi: 10.3766/jaaa.16.9.11. PMID 16515145
- [Background] Saleh HK, Folkeard P, Macpherson E, Scollie S. Adaptation of the Connected Speech Test: Rerecording and Passage Equivalency. Am J Audiol. 2020 Jun 8;29(2):259-264. doi: 10.1044/2019_AJA-19-00052. Epub 2020 Mar 20. PMID 32196353
- [Background] Winkler A, Latzel M, Holube I. Open Versus Closed Hearing-Aid Fittings: A Literature Review of Both Fitting Approaches. Trends Hear. 2016 Feb 15;20:2331216516631741. doi: 10.1177/2331216516631741. PMID 26879562
- [Background] Cox RM, Alexander GC, Gilmore C. Development of the Connected Speech Test (CST). Ear Hear. 1987 Oct;8(5 Suppl):119S-126S. doi: 10.1097/00003446-198710001-00010. PMID 3678650
- [Background] Gabrielsson A, Schenkman BN, Hagerman B. The effects of different frequency responses on sound quality judgments and speech intelligibility. J Speech Hear Res. 1988 Jun;31(2):166-77. doi: 10.1044/jshr.3102.166. PMID 3398490
- [Background] Vasil-Dilaj KA, Cienkowski KM. The influence of receiver size on magnitude of acoustic and perceived measures of occlusion. Am J Audiol. 2011 Jun;20(1):61-8. doi: 10.1044/1059-0889(2010/09-0031). Epub 2011 Jan 28. PMID 21278262

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants With Hearing Loss: Individuals with hearing loss that meet the candidacy to wear hearing aids with various coupling methods. All participants will be exposed to all interventions in a single session
  Recordings of Hearing Aids with Open Domes: Receiver-in-the-Canal hearing aids will be used which are programmed to the participant's hearing loss and will be coupled to open domes. Recordings will be made of hearing aid output on a head and torso simulator and played back to participants over headphones.
  Recordings of Hearing Aids with Closed Domes: Receiver-in-the-Canal hearing aids will be used which are programmed to the participant's hearing loss and will be coupled with closed domes. Recordings will be made of hearing aid output on a head and torso simulator and played back to participants over headphones.
  Recordings of Hearing Aids with Novel State 1: Receiver-in-the-Canal hearing aids will be used which are programmed to the participant's hearing loss and will be coupled with the new coupling method in its first state. Recordings will be made of hearing aid output on a head and torso simulator and played back to participants over headphones.
  Recordings of Hearing Aids with Novel State 2: Receiver-in-the-Canal hearing aids will be used which are programmed to the participant's hearing loss and will be coupled with the new coupling method in its second state. Recordings will be made of hearing aid output on a head and torso simulator and played back to participants over headphones.
Period: Intake and Consent Form Completion
Arm/Group | Participants With Hearing Loss
Started | 20
Completed | 20
Not Completed | 0
Period: Breaks Between Appointment 1 and 2
Arm/Group | Participants With Hearing Loss
Started | 20
Completed | 20
Not Completed | 0
Period: Streaming Sound Quality Task
Arm/Group | Participants With Hearing Loss
Started | 20
Completed | 20
Not Completed | 0
Period: Situational Preference Task
Arm/Group | Participants With Hearing Loss
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Participants With Hearing Loss: All participants will be assessed under all interventions.
  Recordings of Hearing Aids with Open Domes: Receiver-in-the-Canal hearing aids will be used which are programmed to the participant's hearing loss and will be coupled to open domes. Recordings will be made of hearing aid output on a head and torso simulator and played back to participants over headphones.
  Recordings of Hearing Aids with Closed Domes: Receiver-in-the-Canal hearing aids will be used which are programmed to the participant's hearing loss and will be coupled with closed domes. Recordings will be made of hearing aid output on a head and torso simulator and played back to participants over headphones.
  Recordings of Hearing Aids with Novel State 1: Receiver-in-the-Canal hearing aids will be used which are programmed to the participant's hearing loss and will be coupled with the new coupling method in its first state. Recordings will be made of hearing aid output on a head and torso simulator and played back to participants over headphones.
  Recordings of Hearing Aids with Novel State 2: Receiver-in-the-Canal hearing aids will be used which are programmed to the participant's hearing loss and will be coupled with the new coupling method in its second state. Recordings will be made of hearing aid output on a head and torso simulator and played back to participants over headphones.
Arm/Group | Participants With Hearing Loss
Number analyzed (Participants) | 20
Age, Continuous [Mean (Full Range); unit: Years] | 75 [61 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Hearing Thresholds [Mean (Full Range); unit: dB HL (decibel Hearing Loss)] — Hearing thresholds are measured via a hearing test. A hearing test is conducted by a licensed professional who is trained to conduct hearing tests and determine the severity of a participant's hearing loss. Depending on the configuration and severity of the hearing loss dictates if participants meet the requirements to join a clinical study. Hearing thresholds are measured across various frequencies and certain frequencies can differ significantly between participants. The average of four frequencies (500, 1000, 2000, and 4000 Hz (i.e., Pure Tone Average (PTA)) summarizes a participants loss.
  dB HL (decibel Hearing Loss) | 41 [25 to 57.5]
Hearing aid experience [Mean (Full Range); unit: years] | 7.73 [0 to 27]

OUTCOME MEASURES:

1. Primary Outcome: Sound Quality Ratings While Streaming
Description: Hearing aid recordings of different coupling options will be presented via a Multiple Stimuli with Reference and Anchor (MUSHRA) paradigm, where participants will rate and compare sound quality attributes between them.
  Ratings will be made on a scale where 0 would the minimum value and 100 would be the maximum value.
  Fullness: Higher scores indicate that participants found the recording to be fuller (thicker/richer sound). Higher scores indicate a better outcome.
  Sharpness: Higher scores indicate that participants found the recording to be sharper (thinner/more shrill). Lower scores indicate a better outcome.
  Overall Impression: Higher scores indicate that participants had an increased preference towards the recording when compared to the other recordings. Higher scores indicate a better outcome.
Time Frame: 60 minutes
Measure: Mean (Full Range); unit: Units on a rating scale
Groups:
- Sound Quality Ratings: All 20 participants were asked to listen to various recorded stimuli and were asked to rate preference for each stimuli based on certain sound quality attributes (overall impression, sharpness, and fullness).
  All 4 interventions were implemented at once (as is the nature of the MUSHRA) and ratings were made at the same time.
Arm/Group | Sound Quality Ratings
Number analyzed (Participants) | 20
Units on a rating scale
  Open Domes - Pop - Overall Impression | 43.15 [1 to 83]
  Vented Domes - Pop - Overall Impression | 60.025 [17 to 91]
  State 2 - Pop - Overall Impression | 64.025 [34 to 96]
  State 1 - Pop - Overall Impression | 49.00 [11 to 91]
  Open Domes - Speech - Overall Impression | 62.9 [13 to 93]
  Vented Domes - Speech - Overall Impression | 68.325 [35 to 94]
  State 2 - Speech - Overall Impression | 67.575 [30 to 95]
  State 1 - Speech - Overall Impression | 67.65 [23 to 95]
  Open Domes - Classical - Overall Impression | 68.525 [0 to 94]
  Vented Domes - Classical - Overall Impression | 71.775 [35 to 94]
  State 2 - Classical - Overall Impression | 65.725 [35 to 92]
  State 1 - Classical - Overall Impression | 61.525 [31 to 92]
  Open Domes - Pop - Sharpness | 68.175 [23 to 93]
  Vented Domes - Pop - Sharpness | 55.875 [15 to 92]
  State 2 - Pop - Sharpness | 49.725 [7 to 92]
  State 1 - Pop - Sharpness | 57.725 [29 to 88]
  Open Domes - Classical - Sharpness | 61.875 [17 to 95]
  Vented Domes - Classical - Sharpness | 57.1 [3 to 95]
  State 2 - Classical - Sharpness | 61.75 [20 to 95]
  State 1 - Classical - Sharpness | 60.275 [13 to 92]
  Open Domes - Speech - Sharpness | 56.95 [10 to 93]
  Vented Domes - Speech - Sharpness | 46.5 [10 to 96]
  State 2 - Speech - Sharpness | 54.525 [10 to 95]
  State 1 - Speech - Sharpness | 51.275 [12 to 93]
  Open Domes - Pop - Fullness | 45.525 [14 to 90]
  Vented Domes - Pop - Fullness | 61.525 [17 to 95]
  State 2 - Pop - Fullness | 66.55 [11 to 91]
  State 1 - Pop - Fullness | 51.725 [30 to 91]
  Open Domes - Classical - Fullness | 60.8 [0 to 91]
  Vented Domes - Classical - Fullness | 67.125 [28 to 99]
  State 2 - Classical - Fullness | 58.425 [26 to 92]
  State 1 - Classical - Fullness | 59.025 [25 to 91]
  Open Domes - Speech - Fullness | 57.875 [5 to 93]
  Vented Domes - Speech - Fullness | 64.1 [23 to 94]
  State 2 - Speech - Fullness | 60.3 [31 to 93]
  State 1 - Speech - Fullness | 59.875 [29 to 94]

2. Secondary Outcome: Situational Preference Ratings
Description: Hearing aid recordings of different listening situations through different coupling options will be presented via a Multiple Stimuli with Reference and Anchor (MUSHRA) paradigm, where participants will indicate preferences between different recordings.
  Ratings will be made on a scale where 0 would the minimum value and 100 would be the maximum value. Higher scores indicate increased preferred sound quality.
  Higher scores will indicate that participants had an increased preference towards that recording when compared to the other recordings. In this measure, on
Time Frame: 60 Minutes
Population: This is a single arm study, where the arm is participants with hearing loss and who are exposed to multiple interventions (i.e., open domes, closed domes, state 1, and state 2) within-subjects design.
Measure: Mean (Full Range); unit: Units on a rating scale
Groups:
- Sound Quality Ratings - Situational Preference: All 20 participants were asked to listen to various recorded stimuli and were asked to rate overall sound quality
  All 4 interventions were implemented at once (as is the nature of the MUSHRA) and ratings were made at the same time.
Arm/Group | Sound Quality Ratings - Situational Preference
Number analyzed (Participants) | 20
Units on a rating scale
  State 2 - Mic Off - Music - Stream | 82.225 [64 to 100]
  State 2 - Mic On - Music - Stream | 23.125 [2 to 70]
  State 1 - Mic Off - Music - Stream | 50.35 [6 to 99]
  State 1 - Mic On - Music - Stream | 21.95 [2 to 59]
  State 2 - Mic Off - Speech - Stream | 84.225 [9 to 98]
  State 2 - Mic On - Speech - Stream | 29.2 [2 to 72]
  State 1 - Mic Off - Speech - Stream | 63.175 [27 to 98]
  State 1 - Mic On - Speech - Stream | 28.925 [2 to 72]
  State 2 - Mic Off - Music - Noise | 37.6 [1 to 99]
  State 2 - Mic On - Music - Noise | 42.55 [0 to 90]
  State 1 - Mic Off - Music - Noise | 45.90 [10 to 79]
  State 1 - Mic On - Music - Noise | 43.675 [1 to 89]
  State 2 - Mic Off - Speech - Noise | 43.1 [0 to 97]
  State 2 - Mic On - Speech - Noise | 41.675 [2 to 87]
  State 1 - Mic Off - Speech - Noise | 51.225 [5 to 96]
  State 1 - Mic On - Speech - Noise | 39.625 [3 to 73]

ADVERSE EVENTS:
Time Frame: Participants were exposed to multiple interventions at once and had the ability to cycle through the various interventions (frequency curves). For this reason, adverse event data would have been collected per task and not intervention due to the quick exposure to multiple interventions. Adverse Event Data per participant was collected and is reported below. Streaming sound quality task - 60 minutes Situational preference task - 60 minutes
Groups:
- Participants With Hearing Loss - Intake and Consent Form: Participants were recruited to join the study. During recruitment, participants would review and sign the consent form and a hearing test was completed. The same participants then moved on to the next two tasks.
- Participants With Hearing Loss - Streaming Sound Quality Task: All participants will be assessed under all interventions.
  Recordings of Hearing Aids with Open Domes: Receiver-in-the-Canal hearing aids will be used which are programmed to the participant's hearing loss and will be coupled to open domes. Recordings will be made of hearing aid output on a head and torso simulator and played back to participants over headphones.
  Recordings of Hearing Aids with Closed Domes: Receiver-in-the-Canal hearing aids will be used which are programmed to the participant's hearing loss and will be coupled with closed domes. Recordings will be made of hearing aid output on a head and torso simulator and played back to participants over headphones.
  Recordings of Hearing Aids with Novel State 1: Receiver-in-the-Canal hearing aids will be used which are programmed to the participant's hearing loss and will be coupled with the new coupling method in its first state. Recordings will be made of hearing aid output on a head and torso simulator and played back to participants over headphones.
  Recordings of Hearing Aids with Novel State 2: Receiver-in-the-Canal hearing aids will be used which are programmed to the participant's hearing loss and will be coupled with the new coupling method in its second state. Recordings will be made of hearing aid output on a head and torso simulator and played back to participants over headphones.
- Participants With Hearing Loss - Situational Preference Task: All participants will be assessed under all interventions.
  Recordings of Hearing Aids with Novel State 1: Receiver-in-the-Canal hearing aids will be used which are programmed to the participant's hearing loss and will be coupled with the new coupling method in its first state. Recordings will be made of hearing aid output on a head and torso simulator and played back to participants over headphones.
  Recordings of Hearing Aids with Novel State 2: Receiver-in-the-Canal hearing aids will be used which are programmed to the participant's hearing loss and will be coupled with the new coupling method in its second state. Recordings will be made of hearing aid output on a head and torso simulator and played back to participants over headphones.
Arm/Group | Participants With Hearing Loss - Intake and Consent Form | Participants With Hearing Loss - Streaming Sound Quality Task | Participants With Hearing Loss - Situational Preference Task
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-30): https://cdn.clinicaltrials.gov/large-docs/59/NCT05377359/Prot_SAP_000.pdf